CLINICAL TRIAL: NCT07000045
Title: Coronary Calcified Nodule Management With Rotational Atherectomy Plus Shockwave Intravascular Lithotripsy vs. Intravascular Lithotripsy Alone: A Prospective, Randomized Trial (NODULE-SHOCK)
Brief Title: Intravascular Lithotripsy With or Without Rotational Atherectomy for Coronary Calcified Nodule Treatment
Acronym: NODULE-SHOCK
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Annapoorna Kini (Other)
Responsible Party: Sponsor-Investigator, Annapoorna Kini, Professor, Icahn School of Medicine at Mount Sinai
Organization: Icahn School of Medicine at Mount Sinai (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: STUDY-25-00266; ISR20250319 (Other Grant/Funding Number: ShockWave Medical, Inc.)
Record Dates: First submitted 2025-05-23; First posted 2025-05-31 (Actual); Last update posted 2025-10-09 (Actual); Status verified 2025-10

CONDITIONS: Coronary Artery Disease; Coronary Calcification
Keywords: Coronary calcification; Calcified nodule; Intravascular lithotripsy; Rotational atherectomy; Optical coherence tomography; Percutaneous coronary intervention
MeSH Terms: conditions — Coronary Artery Disease | interventions — Atherectomy, Coronary

STUDY DESIGN:
Intervention Model Description: Cohort A: RA + IVL vs IVL alone for calcified nodules Cohort B: Operator-determined IVL pulses vs Maximum IVL pulses for non-CN severe calcium
Who Masked: Participant
Masking Description: Participants are blinded to treatment allocation. Operators and investigators are unblinded.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (4):
- RA + IVL (Cohort A) (Experimental): Patients with coronary calcified nodules treated with rotational atherectomy followed by intravascular lithotripsy for lesion preparation prior to stenting.
  Interventions: Device: Intravascular lithotripsy; Device: Rotational atherectomy
- IVL alone (Cohort A) (Active Comparator): Patients with coronary calcified nodules treated with intravascular lithotripsy alone for lesion preparation prior to stenting.
  Interventions: Device: Intravascular lithotripsy
- Maximum IVL pulses (Cohort B) (Experimental): Patients with non-nodular severe coronary calcium treated with intravascular lithotripsy prior to stenting using the maximum number of pulses per manufacturer's instructions.
  Interventions: Device: Intravascular lithotripsy
- Operator-determined IVL pulses (Cohort B) (Active Comparator): Patients with non-nodular severe coronary calcium treated with intravascular lithotripsy prior to stenting using a pulse number determined at the operator's discretion.
  Interventions: Device: Intravascular lithotripsy

INTERVENTIONS:
Device: Intravascular lithotripsy — Intravascular lithotripsy device used for calcium modification in coronary lesions, using either operator-determined or maximum pulsed numbers for lesion preparation prior to stenting.
Device: Rotational atherectomy — Rotational atherectomy device used to debulk calcified nodules before IVL and stent implantation.
  Arms: RA + IVL (Cohort A)

SUMMARY:
The NODULE-SHOCK trial is a prospective, investigator-initiated, single-center, randomized controlled trial designed to compare the efficacy of intravascular lithotripsy (IVL) with or without rotational atherectomy (RA) in patients with coronary calcified nodules (Cohort A), and operator-determined vs maximum IVL pulses in patients with non-nodular severe coronary calcium (Cohort B).

DETAILED DESCRIPTION:
The trial consists of two cohorts:

* Patients with calcified nodules (CN) (Cohort A)
* Patients with non-nodular severe coronary calcium (Cohort B)

Randomization will occur as follows:

* Rotational atherectomy followed by intravascular lithotripsy (IVL) or IVL alone for lesion preparation prior to stenting (Cohort A).
* Operator-determined or maximum IVL pulses prior to stenting. (Cohort B)

The trial is designed to compare two calcium modification strategies in each cohort with regard to the primary endpoints of post-procedural minimum stent area assessed by optical coherence tomography at the CN site (Cohort A) and at the site of maximum calcification (Cohort B).

ELIGIBILITY:
Inclusion Criteria

* Age ≥18 years who signed written informed consent
* Presence of a clinical indication for coronary intervention
* Patients undergoing PCI for a de novo calcified lesion with planned drug-eluting stent (DES) implantation
* Native coronary artery with significant stenosis defined as:
* ≥70% and <100% stenosis on angiography, or
* 50-70% stenosis with evidence of ischemia (positive stress test, FFR ≤ 0.8, or OCT minimal lumen area (MLA) ≤ 4.0 mm2)
* Reference vessel diameter: ≥2.5 mm to ≤ 4.0 mm
* Lesion length: ≥5mm
* Moderate to severe calcification of the target lesion confirmed by angiography
* Thrombolysis in Myocardial Infarction (TIMI) flow grade 3 at baseline

Exclusion Criteria

* Cardiogenic shock at the time of procedure
* Primary PCI for ST-segment elevation myocardial infarction (STEMI)
* Pregnant, nursing, or childbearing potential without adequate contraception
* Known allergy or contraindication to DAPT (aspirin, clopidogrel, prasugrel, ticagrelor)
* Planned surgery within 6 months unless DAPT can be maintained
* Life expectancy <12 months due to a serious medical illness (e.g., advanced cancer, end-stage heart failure)
* Severe kidney dysfunction (CrCl <30 mL/min) without dialysis
* Concurrent participation in another investigational study
* Referral for coronary artery bypass grafting (CABG) after a heart team discussion
* Angiographic evidence of thrombus at the target lesion
* Angiographic evidence of significant dissection at the treatment site prior to intervention
* Lesion with a previously placed stent within 10mm (visual estimate)
* Last remaining vessel with severely compromised left ventricular function (LVEF <30%)
* Target lesion within a saphenous vein graft (SVG)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2025-10-06 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Minimum stent area (MSA) | Immediately after Index procedure
  Post-procedural minimum stent area measured at the site of the calcified nodule (Cohort A) or the point of maximum calcification (Cohort B), as assessed by optical coherence tomography (OCT)

SECONDARY OUTCOMES:
Number of Calcium fractures | Immediately after Index procedure
  Number and presence of post-IVL calcium fractures identified on OCT
Target vessel failure (TVF) | during hospitalization, approximately 1-2 days, 30 days, and 12 months
  Target vessel failure (TVF) defined as composite of cardiac death, target vessel myocardial infarction, and target vessel revascularization
Stent thrombosis | 12 months
  Definite or probable stent thrombosis according to academic research consortium-2 (ARC-2) definitions.
  Definite stent thrombosis is defined as the presence of a thrombus within the stent, within 5 mm of the stent edge, or in a side branch of the stented segment, confirmed by angiography or pathology, along with evidence of acute ischemia such as symptoms, ECG changes, or elevated cardiac biomarkers.
  Probable is defined as a myocardial infarction in the territory of the stented vessel without angiographic confirmation and without another obvious cause.
Device success | Immediately after Index procedure
  Successful lesion crossing and device delivery to the target site
Angiographic success | Immediately after Index procedure
  Angiographic success defined as stent deployment with residual stenosis <30% and TIMI 3 flow without significant angiographic complications (perforation, major dissection, distal embolization, slow flow, or no flow)
Procedural success | Immediately after Index procedure
  Procedural success defined as angiographic success and no in-hospital TVF
Bailout or adjunctive calcium modification | Intraoperatively during Index procedure
  Use of additional calcium modification device beyond initial randomized strategy
Pre- and post-dilatation ballon size | Immediately before and after Index procedure
  Balloon size recorded during lesion preparation and post-dilatation
Pre- and post-dilatation inflation pressure | Immediately before and after Index procedure
  Inflation pressure recorded during lesion preparation and post-dilatation
Total number of IVL pulses delivered to the lesion during treatment | Intraoperatively during Index procedure
  IVL pulse characteristics - Total number of IVL pulses delivered to the lesion during treatment relative to overall lesion length and calcified segment length
Lesion length of IVL pulses delivered | Intraoperatively during Index procedure
  IVL pulse characteristics - The lesion length over which pulses were applied, relative to overall lesion length and calcified segment length

CONTACTS AND LOCATIONS:
Overall Officials: Annapoorna S Kini, MD, Principal Investigator — Icahn School of Medicine at Mount Sinai
Locations (1):
- Mount Sinai Hospital, New York, New York, United States

IPD SHARING:
Plan to Share IPD: No
De-identified data will only be shared with the study funder for internal use. No public IPD sharing is planned.